CLINICAL TRIAL: NCT01838655
Title: A Pilot Study of Nitisinone in the Treatment of Oculocutaneous Albinism, Type 1B
Brief Title: Nitisinone for Type 1B Oculocutaneous Albinism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130124; 13-EI-0124 (Other: NIH Combined NeuroScience Institutional Review Board)
Record Dates: First submitted 2013-04-20; First posted 2013-04-24 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2017-10

CONDITIONS: Albinism; Vision Loss
Keywords: Albinism; Nitisinone; Melanin; Vision Loss
MeSH Terms: conditions — Albinism; Vision Disorders | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitisinone (Experimental): Oral administration of nitisinone
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — Oral dose of 2mg daily for 12 months.
  Other Names: Orfadin

SUMMARY:
Background:

- Oculocutaneous albinism, type 1B (OCA1B) is a genetic disease caused by problems in the gene that makes tyrosine. Tyrosine is an amino acid needed to produce pigment in the skin, hair, and eyes. People with OCA1B have pale skin, white hair, and light-colored eyes. Pigment in the back of the eye helps vision, so people with OCA-1B often have visual problems. Researchers want to see if a drug called nitisinone can help improve eye pigmentation and vision in people with OCA1B. Nitisinone is approved for treating a related genetic disease that causes problems with tyrosine, so it may help people with OCA1B.

Objectives:

- To see if nitisinone can help improve eye pigmentation and vision in people with OCA1B.

Eligibility:

- Individuals at least 18 years of age who have OCA1B.

Design:

* This study will last about 18 months. It requires eight outpatient visits, each about 3 months apart. Each visit will require 1 to 2 days of testing.
* Participants will be screened with a physical exam, eye exam, and medical history. They will have additional vision and neurological tests. They will be tested to see how their brain and retinas respond to light. They will also take hair and blood samples, and answer questions about diet.
* Participants will receive the study drug. They will take one pill a day for 1 year. They will keep track of the dose in a study diary.
* At the outpatient visits, participants will have the following tests:
* Medical history and physical exam
* Neurological and eye exams
* Retina function tests
* Tests of the skin and brain's response to light
* Blood and urine tests
* Dietary consultation
* Visual function questionnaire.
* After the end of the study, participants will return to the care of their regular eye doctor.

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to evaluate oral nitisinone as a treatment that improves ocular pigmentation in adult participants with oculocutaneous albinism, type 1B (OCA1B). Secondary objectives of this study are to determine whether the selected outcome measures are robust enough to use in a larger trial and to assess whether oral nitisinone improves visual function, skin pigmentation, and hair pigmentation in participants with OCA1B.

Study Population: Five participants with OCA1B will be enrolled initially. However, up to an additional three participants may be enrolled to account for participants who withdraw from the study for any reason before the Month 12 visit.

Design: In this pilot, phase 1/2, single-site, prospective, open label trial, participants will receive 2 mg of oral nitisinone daily for at least one year, and they will be followed for at least 18 months. Ocular and non-ocular data will be collected at least every three months, with the first follow-up visit occurring three months after the final baseline visit. Participants will be required to have at least 8 outpatient visits at the NEI clinic over a period of 18 months. This study has a common termination date and therefore may continue for up to four years.

Outcome Measures: The primary outcome for the study is the absolute mean change in iris pigmentation on an 8-point scale at 12 months as compared to baseline. Participants left and right eyes will be analyzed. The absolute mean change in iris pigmentation for each eye on an 8-point scale at 3, 6 and 9 months compared to baseline will be assessed as secondary outcomes. Other secondary outcomes include the absolute and percent change in semi-quantitative iris pigmentation on image analysis; the absolute change in electronic visual acuity (EVA) for each eye and binocular vision; the absolute change in contrast sensitivity without glare, with medium glare, and with high glare for binocular vision; the absolute change in full-field ERG measures for each eye; and the absolute and percent change in melanin content in skin using skin reflectometry at 3, 6, 9 and 12 months as compared to baseline; Qualitative changes in hair, skin, and fundus pigmentation at 3, 6, 9 and 12 months as compared to previous visit will be assessed. The absolute and percent change in hair melanin will also be assessed at 12 months as compared to baseline. The number and severity of adverse events and the number of withdrawals will be assessed as safety outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, when applicable.

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol s informed consent document.
3. Participant must have normal renal function, liver function, and platelet counts or have mild abnormalities no greater than grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
4. Any female participant of childbearing potential must have a negative pregnancy test at screening and must be willing to undergo pregnancy testing immediately prior to the start of the investigational product and while on the investigational product.
5. Any female participant of childbearing potential and any male participant able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse, or must agree to practice two effective methods of contraception while taking the investigational product and for at least two months following the last dose of investigational product. Acceptable methods of contraception include:

   * Hormonal contraception (i.e., birth control pills, injected hormones, dermal patch, or vaginal ring),
   * Intrauterine device,
   * Barrier methods (diaphragm, condom) with spermicide, or
   * Surgical sterilization (tubal ligation).
6. Participant must have OCA1B, as defined by ALL (a-d) of the following criteria:

   1. Participant has ophthalmic signs or symptoms of albinism, including:

      * Bilateral visual acuity E-ETDRS EVA letter score of less than or equal to 83 (i.e., Snellen equivalent of 20/25 or worse) that is not attributable to any other pathology.
      * Bilateral iris transillumination that can be seen in clinical photographs.
   2. Predominant contralateral decussation of ganglion cell axons, as determined by pattern visual evoked potential (VEP).
   3. Participant has at least one definitive mutation in the OCA1 gene (tyrosinase).
   4. Participant has no definitive mutations in the OCA2 gene.

EXCLUSION CRITERIA:

* Participant is pregnant or breast-feeding.
* Participant is a male AND has a definitive mutation in the OA1 gene.
* Participant has any of the following abnormal laboratory test results:

  1. Serum potassium < 3.0 mEq/L,
  2. Serum CK > 500 U/L,
  3. Hemoglobin < 10.0 g/dL,
  4. White blood cell (WBC) count < 3.0 k/microL,
  5. Plasma tyrosine > 150 microM,
  6. ESR > 100 mm/h, and/or
  7. Serum T4 > 15 microg/dL OR Serum T4 < 4 microg/dL.
* Participant has keratopathy.
* Participant has a current malignancy.
* Participant has open skin lesions.
* Participant is on a diet that deliberately increases protein intake to disproportionate levels (e.g., Atkins diet). The diet must be reasonably balanced, as determined by a dietician.
* Participant has uncontrolled hypertension, defined as systolic blood pressure above 180 mmHg or diastolic blood pressure above 95 mmHg.
* Participant has another chronic ocular disease that may confound the results of visual tests, such as age-related macular degeneration, cataract of possible visual significance, or uncontrolled glaucoma.
* Participant drinks more than the equivalent of two glasses of wine per day on average, has a history of alcohol abuse, or has a severe liver illness.
* Participant s liver is > 3 cm below the right costal margin.
* Participant has a muscle disease.
* Participant is currently taking a medication known to cause elevated liver function tests including statins/HMG-Co-A reductase inhibitors (e.g., lovastatin, simvastatin); anti-epileptic medications (e.g., carbamazepine, phenytoin, phenobarbital); tetracycline or its derivatives, if used chronically; acetaminophen, if used daily/chronically; amiodarone; and any other medications with known significant liver toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04-16; Primary Completion 2016-07-11 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hertle RW, Anninger W, Yang D, Shatnawi R, Hill VM. Effects of extraocular muscle surgery on 15 patients with oculo-cutaneous albinism (OCA) and infantile nystagmus syndrome (INS). Am J Ophthalmol. 2004 Dec;138(6):978-87. doi: 10.1016/j.ajo.2004.07.029. PMID 15629289
- [Background] Giebel LB, Tripathi RK, King RA, Spritz RA. A tyrosinase gene missense mutation in temperature-sensitive type I oculocutaneous albinism. A human homologue to the Siamese cat and the Himalayan mouse. J Clin Invest. 1991 Mar;87(3):1119-22. doi: 10.1172/JCI115075. PMID 1900309
- [Background] Giebel LB, Tripathi RK, Strunk KM, Hanifin JM, Jackson CE, King RA, Spritz RA. Tyrosinase gene mutations associated with type IB ("yellow") oculocutaneous albinism. Am J Hum Genet. 1991 Jun;48(6):1159-67. PMID 1903591
- [Result] Adams DR, Menezes S, Jauregui R, Valivullah ZM, Power B, Abraham M, Jeffrey BG, Garced A, Alur RP, Cunningham D, Wiggs E, Merideth MA, Chiang PW, Bernstein S, Ito S, Wakamatsu K, Jack RM, Introne WJ, Gahl WA, Brooks BP. One-year pilot study on the effects of nitisinone on melanin in patients with OCA-1B. JCI Insight. 2019 Jan 24;4(2):e124387. doi: 10.1172/jci.insight.124387. PMID 30674731
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-EI-0124.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants with OCA1B will be enrolled initially. However, up to an additional three participants may be enrolled to account for participants who withdraw from the study for any reason before the Month 12 visit.
Period: Overall Study
Arm/Group | Nitisinone
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 38.8 [24 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Mean Change in Iris Pigmentation on an 8-point Iris Transillumination Scale at 12 Months as Compared to Baseline. Participants Left and Right Eyes Will be Analyzed.
Description: High-resolution (2544x1696) digital images of the anterior segment of both eyes were captured prior to pupil dilation using diffuse illumination and iris transillumination. An independent reviewer selected two transillumination images from each eye of each participant for each visit according to preset quality criteria. Images were coded, randomized and presented to a panel of 18 graders on a SHARP 90" HD LED TV. After instruction and a practice dataset, graders scored each image using an 8-point scale. Graders could score images with a single decimal place if they felt an image fell in between two of the standards. The iris transillumination scale ranged from 0 to 8, with lower scores reflective of greater iris pigmentation (melanin content). The mean across all graders and the two images for each participant's eye at baseline and 12 months was calculated; these mean grades were then used to calculate absolute change from baseline at 12 months.
Time Frame: Baseline and 12 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 1.2 (1.68)
  OS: number analyzed (eyes) | 5
  OS | 0.9 (1.52)

2. Secondary Outcome: Absolute Mean Change in Iris Pigmentation on an 8-point Iris Transillumination Scale at 3 Months as Compared to Baseline. Participants Left and Right Eyes Will be Analyzed.
Description: High-resolution (2544x1696) digital images of the anterior segment of both eyes were captured prior to pupil dilation using diffuse illumination and iris transillumination. An independent reviewer selected two transillumination images from each eye of each participant for each visit according to preset quality criteria. Images were coded, randomized and presented to a panel of 18 graders on a SHARP 90" HD LED TV. After instruction and a practice dataset, graders scored each image using an 8-point scale. Graders could score images with a single decimal place if they felt an image fell in between two of the standards. The iris transillumination scale ranged from 0 to 8, with lower scores reflective of greater iris pigmentation (melanin content). The mean across all graders and the two images for each participant's eye at baseline and 3 months was calculated; these mean grades were then used to calculate absolute change from baseline at 3 months.
Time Frame: Baseline and 3 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 0.8 (1.04)
  OS: number analyzed (eyes) | 5
  OS | 0.9 (1.23)

3. Secondary Outcome: Absolute Mean Change in Iris Pigmentation on an 8-point Iris Transillumination Scale at 6 Months as Compared to Baseline. Participants Left and Right Eyes Will be Analyzed.
Description: High-resolution (2544x1696) digital images of the anterior segment of both eyes were captured prior to pupil dilation using diffuse illumination and iris transillumination. An independent reviewer selected two transillumination images from each eye of each participant for each visit according to preset quality criteria. Images were coded, randomized and presented to a panel of 18 graders on a SHARP 90" HD LED TV. After instruction and a practice dataset, graders scored each image using an 8-point scale. Graders could score images with a single decimal place if they felt an image fell in between two of the standards. The iris transillumination scale ranged from 0 to 8, with lower scores reflective of greater iris pigmentation (melanin content). The mean across all graders and the two images for each participant's eye at baseline and 6 months was calculated; these mean grades were then used to calculate absolute change from baseline at 6 months.
Time Frame: Baseline and 6 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 0.6 (0.39)
  OS: number analyzed (eyes) | 5
  OS | 0.4 (0.31)

4. Secondary Outcome: Absolute Mean Change in Iris Pigmentation on an 8-point Iris Transillumination Scale at 9 Months as Compared to Baseline. Participants Left and Right Eyes Will be Analyzed.
Description: High-resolution (2544x1696) digital images of the anterior segment of both eyes were captured prior to pupil dilation using diffuse illumination and iris transillumination. An independent reviewer selected two transillumination images from each eye of each participant for each visit according to preset quality criteria. Images were coded, randomized and presented to a panel of 18 graders on a SHARP 90" HD LED TV. After instruction and a practice dataset, graders scored each image using an 8-point scale. Graders could score images with a single decimal place if they felt an image fell in between two of the standards. The iris transillumination scale ranged from 0 to 8, with lower scores reflective of greater iris pigmentation (melanin content). The mean across all graders and the two images for each participant's eye at baseline and 9 months was calculated; these mean grades were then used to calculate absolute change from baseline at 9 months.
Time Frame: Baseline and 9 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 0.9 (1.06)
  OS: number analyzed (eyes) | 5
  OS | 0.6 (0.60)

5. Secondary Outcome: Absolute Change in Semi-quantitative Iris Pigmentation for Each Eye at 3 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 3 months; these mean grades were then used to calculate absolute change from baseline.
Time Frame: Baseline and 3 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 1.2 (1.04)
  OS: number analyzed (eyes) | 5
  OS | 0.6 (0.82)

6. Secondary Outcome: Absolute Change in Semi-quantitative Iris Pigmentation for Each Eye at 6 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 6 months; these mean grades were then used to calculate absolute change from baseline.
Time Frame: Baseline and 6 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 0.4 (0.55)
  OS: number analyzed (eyes) | 5
  OS | 0.1 (0.22)

7. Secondary Outcome: Absolute Change in Semi-quantitative Iris Pigmentation for Each Eye at 9 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 9 months; these mean grades were then used to calculate absolute change from baseline.
Time Frame: Baseline and 9 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 0.8 (0.76)
  OS: number analyzed (eyes) | 5
  OS | 0.7 (0.84)

8. Secondary Outcome: Absolute Change in Semi-quantitative Iris Pigmentation for Each Eye at 12 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 12 months; these mean grades were then used to calculate absolute change from baseline.
Time Frame: Baseline and 12 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
scores on a scale
  OD: number analyzed (eyes) | 5
  OD | 1.4 (1.39)
  OS: number analyzed (eyes) | 5
  OS | 1.2 (1.15)

9. Secondary Outcome: Percent Change in Semi-quantitative Iris Pigmentation for Each Eye at 3 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 3 months; these mean grades were then used to calculate percentage change from baseline.
Time Frame: Baseline and 3 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
percentage change
  OD: number analyzed (eyes) | 5
  OD | 66.7 (51.37)
  OS: number analyzed (eyes) | 5
  OS | 29.0 (41.29)

10. Secondary Outcome: Percent Change in Semi-quantitative Iris Pigmentation for Each Eye at 6 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 6 months; these mean grades were then used to calculate percentage change from baseline.
Time Frame: Baseline and 6 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
percentage change
  OD: number analyzed (eyes) | 5
  OD | 23.3 (32.49)
  OS: number analyzed (eyes) | 5
  OS | 4.0 (8.94)

11. Secondary Outcome: Percent Change in Semi-quantitative Iris Pigmentation for Each Eye at 9 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 9 months; these mean grades were then used to calculate percentage change from baseline.
Time Frame: Baseline and 9 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
percentage change
  OD: number analyzed (eyes) | 5
  OD | 42.0 (42.66)
  OS: number analyzed (eyes) | 5
  OS | 34.0 (42.19)

12. Secondary Outcome: Percent Change in Semi-quantitative Iris Pigmentation for Each Eye at 12 Months as Compared to Baseline
Description: In Adobe Photoshop 7.0 the high resolution slit lamp image was divided into 4 quadrants with vertical and horizontal lines transecting the center of the iris. Using the elliptical marquee tool, a circle, approximately 0.25 times the diameter of the iris, was drawn in the center of each quadrant. Gaussian blur with radius of 50 was applied to the area enclosed in the 4 circles. With the dropper tool, the red pigment value corresponding to the degree of iris transillumination was sampled at the center of each circle. The 4 values were averaged to yield a composite transillumination score for each subject. Quantified values were then correlated to a scale score from 1 to 8 to generate an 8-point iris transillumination scale, with lower scores reflective of greater iris pigmentation (melanin content). The mean score across the 2 images for each participant's eye was calculated at baseline and 12 months; these mean grades were then used to calculate percentage change from baseline.
Time Frame: Baseline and 12 months
Population: Right (OD) and left (OS) eyes
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
percentage change
  OD: number analyzed (eyes) | 5
  OD | 77.7 (91.94)
  OS: number analyzed (eyes) | 5
  OS | 67.0 (59.75)

13. Secondary Outcome: Absolute Change in Electronic Visual Acuity at 3 Months Compared to Baseline
Description: Visual acuity was measured using the Electronic ETDRS Visual Acuity Testing protocol. Acuity is measured as letters read using an electronic ETDRS program.
Time Frame: Baseline and 3 months
Population: Right (OD) and Left (OS) eyes
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
ETDRS letters
  OD: number analyzed (eyes) | 5
  OD | 1.8 (0.84)
  OS: number analyzed (eyes) | 5
  OS | 6.0 (3.61)

14. Secondary Outcome: Absolute Change in Electronic Visual Acuity at 6 Months Compared to Baseline
Description: as for outcome 13
Time Frame: Baseline and 6 months
Population: Right (OD) and Left (OS) eyes
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
ETDRS letters
  OD: number analyzed (eyes) | 5
  OD | 4.2 (2.17)
  OS: number analyzed (eyes) | 5
  OS | 4.8 (3.42)

15. Secondary Outcome: Absolute Change in Electronic Visual Acuity at 9 Months Compared to Baseline
Description: as for outcome 13
Time Frame: Baseline and 9 months
Population: Right (OD) and Left (OS) eyes
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
ETDRS letters
  OD: number analyzed (eyes) | 5
  OD | 2.8 (2.95)
  OS: number analyzed (eyes) | 5
  OS | 5.6 (2.51)

16. Secondary Outcome: Absolute Change in Electronic Visual Acuity at 12 Months Compared to Baseline
Description: as for outcome 13
Time Frame: Baseline and 12 months
Population: Right (OD) and Left (OS) eyes
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
ETDRS letters
  OD: number analyzed (eyes) | 5
  OD | 5.4 (3.78)
  OS: number analyzed (eyes) | 5
  OS | 5.0 (5.70)

17. Secondary Outcome: Absolute Change in Contrast Sensitivity Without Glare at 3 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. The minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity without glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 3 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.6 (1.52)
  Frequency 3 | 0.8 (0.84)
  Frequency 6 | 0.4 (0.55)
  Frequency 12 | 1.2 (2.17)
  Frequency 18 | 0.6 (1.34)

18. Secondary Outcome: Absolute Change in Contrast Sensitivity Without Glare at 6 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. The minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity without glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 6 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 2.0 (2.83)
  Frequency 3 | 0.2 (0.45)
  Frequency 6 | 1.6 (1.52)
  Frequency 12 | 2.8 (2.95)
  Frequency 18 | 0.0 (0.00)

19. Secondary Outcome: Absolute Change in Contrast Sensitivity Without Glare at 9 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. The minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity without glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 9 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.8 (2.49)
  Frequency 3 | 0.6 (0.55)
  Frequency 6 | 1.0 (1.00)
  Frequency 12 | 1.4 (2.19)
  Frequency 18 | 0.0 (0.00)

20. Secondary Outcome: Absolute Change in Contrast Sensitivity Without Glare at 12 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. The minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity without glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 12 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 2.4 (2.51)
  Frequency 3 | 2.0 (2.55)
  Frequency 6 | 1.8 (1.92)
  Frequency 12 | 1.6 (2.19)
  Frequency 18 | 0.6 (1.34)

21. Secondary Outcome: Absolute Change in Contrast Sensitivity With Medium Glare at 3 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with medium glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 3 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.4 (1.14)
  Frequency 3 | 0.4 (0.55)
  Frequency 6 | 3.6 (3.78)
  Frequency 12 | 0.2 (0.45)
  Frequency 18 | 0.6 (1.34)

22. Secondary Outcome: Absolute Change in Contrast Sensitivity With Medium Glare at 6 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with medium glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 6 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 2.4 (2.88)
  Frequency 3 | 1.4 (1.67)
  Frequency 6 | 1.8 (1.79)
  Frequency 12 | 0.4 (0.89)
  Frequency 18 | 0.6 (1.34)

23. Secondary Outcome: Absolute Change in Contrast Sensitivity With Medium Glare at 9 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with medium glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 9 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 2.0 (2.35)
  Frequency 3 | 1.2 (0.84)
  Frequency 6 | 1.0 (1.00)
  Frequency 12 | 0.6 (1.34)
  Frequency 18 | 0.8 (1.30)

24. Secondary Outcome: Absolute Change in Contrast Sensitivity With Medium Glare at 12 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with medium glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 12 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.4 (2.61)
  Frequency 3 | 1.8 (1.79)
  Frequency 6 | 2.6 (2.79)
  Frequency 12 | 0.4 (0.89)
  Frequency 18 | 1.2 (1.64)

25. Secondary Outcome: Absolute Change in Contrast Sensitivity With High Glare at 3 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with high glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 3 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.2 (1.10)
  Frequency 3 | 1.8 (2.49)
  Frequency 6 | 0.2 (0.45)
  Frequency 12 | 0.2 (0.45)
  Frequency 18 | 0.0 (0.00)

26. Secondary Outcome: Absolute Change in Contrast Sensitivity With High Glare at 6 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with high glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 6 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.0 (1.00)
  Frequency 3 | 1.6 (1.67)
  Frequency 6 | 1.2 (2.17)
  Frequency 12 | 0.4 (0.55)
  Frequency 18 | 0.0 (0.00)

27. Secondary Outcome: Absolute Change in Contrast Sensitivity With High Glare at 9 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with high glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 9 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.4 (0.55)
  Frequency 3 | 0.6 (0.55)
  Frequency 6 | 1.0 (2.24)
  Frequency 12 | 1.6 (2.61)
  Frequency 18 | 0.6 (1.34)

28. Secondary Outcome: Absolute Change in Contrast Sensitivity With High Glare at 12 Months Compared to Baseline
Description: Gratings, images with alternating light and dark bars, assess contrast sensitivity via spatial frequency and contrast. Spatial frequency (SF), the number of pairs of bars (1 light, 1 dark) imaged within a given distance of the retina, is measured as the number of cycles per degree (cpd) of visual angle, where a cycle is 1 pair of bars. Grating of high SF corresponds to narrow bars; grating of low SF corresponds to wide bars. Contrast is the intensity difference between light and dark bars. Minimum contrast required to detect a given SF is the threshold contrast. The lower the threshold contrast, higher the contrast sensitivity. Contrast sensitivity with high glare was measured at frequencies of 1.5, 3, 6, 12, 18 cpd. Absolute change from baseline to 12 months was calculated. Raw values were used for the planned descriptive analysis; logarithmic transformation was not used as formal statistical analysis was not planned and was not appropriate as a majority of the raw values were 0.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
units
  Frequency 1.5 | 1.6 (1.52)
  Frequency 3 | 2.2 (2.28)
  Frequency 6 | 2.6 (3.21)
  Frequency 12 | 1.8 (1.79)
  Frequency 18 | 0.0 (0.00)

29. Secondary Outcome: Absolute Change in Adjusted Melanin Index at 3 Months Compared to Baseline
Description: Microflash 200D is a diffuse reflectance spectrophotometer that uses a prism photodiode to provide information at 10 nm increments along the visual spectrum from 400 to 700 nm. Percent reflectance (PR) at a specific wavelength was placed into context by relating it to the reflectance of a blank at the equivalent wavelength (i.e. relating the object's reflectance to the maximum reflectance possible). Apparent absorbance (AA) at a given wavelength was determined as log10 (PR of blank/PR of object) at that wavelength. Adjusted Melanin (AM) index is calculated as the slope of AA levels from 650 to 700 nm. Lower values of AM index correspond to higher melanin concentrations. Measurements were collected 5 times at each visit from each of the following sites: forehead, inner forearm, outer forearm, inner bicep and lower back. The mean of these five measurements was calculated at each visit. Absolute change from baseline was calculated using these mean values.
Time Frame: Baseline and 3 Months
Measure: Mean (Standard Deviation); unit: Adjusted Melanin Index*10^-5
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Adjusted Melanin Index*10^-5
  Forehead | 16.4 (14.95)
  Inner Bicep | 4.8 (5.24)
  Lower Back | 20.9 (18.91)
  Inner Forearm | 10.7 (5.52)
  Outer Forearm | 10.6 (5.60)

30. Secondary Outcome: Absolute Change in Adjusted Melanin Index at 6 Months Compared to Baseline
Description: as for outcome 29
Time Frame: Baseline and 6 Months
Population: Participant 005 did not have skin reflectometry measurements for any site at Month 6.
Measure: Mean (Standard Deviation); unit: Adjusted Melanin Index*10^-5
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Adjusted Melanin Index*10^-5
  Forehead | 11.8 (4.57)
  Inner Bicep | 8.2 (6.19)
  Lower Back | 9.3 (7.60)
  Inner Forearm | 12.1 (10.59)
  Outer Forearm | 12.6 (6.71)

31. Secondary Outcome: Absolute Change in Adjusted Melanin Index at 9 Months Compared to Baseline
Description: as for outcome 29
Time Frame: Baseline and 9 Months
Population: Participant 002 did not have any skin reflectometry measurements for any site at Month 9.
Measure: Mean (Standard Deviation); unit: Adjusted Melanin Index*10^-5
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Adjusted Melanin Index*10^-5
  Forehead | 10.3 (13.41)
  Inner Bicep | 9.4 (5.85)
  Lower Back | 5.5 (4.12)
  Inner Forearm | 11.6 (7.82)
  Outer Forearm | 1.5 (0.98)

32. Secondary Outcome: Absolute Change in Adjusted Melanin Index at 12 Months Compared to Baseline
Description: as for outcome 29
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: Adjusted Melanin Index*10^-5
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Adjusted Melanin Index*10^-5
  Forehead | 8.3 (6.89)
  Inner Bicep | 7.0 (7.74)
  Lower Back | 4.2 (3.18)
  Inner Forearm | 6.8 (4.20)
  Outer Forearm | 8.6 (5.09)

33. Secondary Outcome: Percent Change in Adjusted Melanin Index at 3 Months Compared to Baseline
Description: Microflash 200D is a diffuse reflectance spectrophotometer that uses a prism photodiode to provide information at 10 nm increments along the visual spectrum from 400 to 700 nm. Percent reflectance (PR) at a specific wavelength was placed into context by relating it to the reflectance of a blank at the equivalent wavelength (i.e. relating the object's reflectance to the maximum reflectance possible). Apparent absorbance (AA) at a given wavelength was determined as log10 (PR of blank/PR of object) at that wavelength. Adjusted Melanin (AM) index is calculated as the slope of AA levels from 650 to 700 nm. Lower values of AM index correspond to higher melanin concentrations. Measurements were collected 5 times at each visit from each of the following sites: forehead, inner forearm, outer forearm, inner bicep and lower back. The mean of these five measurements was calculated at each visit. Percent change from baseline was calculated using these mean values.
Time Frame: Baseline and 3 Months
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Percentage change
  Forehead | 50.1 (49.48)
  Inner Bicep | 40.1 (35.76)
  Lower Back | 201.0 (321.19)
  Inner Forearm | 83.3 (70.69)
  Outer Forearm | 42.1 (22.67)

34. Secondary Outcome: Percent Change in Adjusted Melanin Index at 6 Months Compared to Baseline
Description: as for outcome 33
Time Frame: Baseline and 6 Months
Population: Participant 005 did not have skin reflectometry measurements for any site at Month 6.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Percentage change
  Forehead | 35.4 (14.10)
  Inner Bicep | 123.0 (113.41)
  Lower Back | 117.4 (120.5)
  Inner Forearm | 91.1 (116.26)
  Outer Forearm | 67.9 (56.49)

35. Secondary Outcome: Percent Change in Adjusted Melanin Index at 9 Months Compared to Baseline
Description: as for outcome 33
Time Frame: Baseline and 9 Months
Population: Participant 002 did not have skin reflectometry measurements for any site at Month 9.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Percentage change
  Forehead | 33.2 (44.21)
  Inner Bicep | 94.5 (60.03)
  Lower Back | 39.6 (42.36)
  Inner Forearm | 81.0 (93.51)
  Outer Forearm | 6.0 (5.86)

36. Secondary Outcome: Percent Change in Adjusted Melanin Index at 12 Months Compared to Baseline
Description: as for outcome 33
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Percentage change
  Forehead | 24.7 (21.76)
  Inner Bicep | 104.5 (132.61)
  Lower Back | 32.7 (31.81)
  Inner Forearm | 47.4 (48.10)
  Outer Forearm | 30.5 (7.60)

37. Secondary Outcome: Absolute Change in Melanin Index at 3 Months Compared to Baseline
Description: Microflash 200D is a diffuse reflectance spectrophotometer that uses a prism photodiode to provide information at 10 nm increments along the visual spectrum from 400 to 700 nm. Percent reflectance (PR) at a specific wavelength was placed into context by relating it to the reflectance of a blank at the equivalent wavelength (i.e. relating the object's reflectance to the maximum reflectance possible). Melanin (M) index was calculated as follows:
  Eqn 1= [ (PR at 650nm + PR at 660nm + 0.5*PR at 640nm + 0.5*PR at 670nm)/3 ]/100; M index = 100*log (1/Eqn 1) Higher values of M index correspond to higher melanin concentrations. Measurements were collected 5 times at each visit from each of the following sites:forehead, inner forearm, outer forearm, inner bicep and lower back. The mean of these five measurements was calculated at each visit. Absolute change from baseline was calculated using these mean values.
Time Frame: Baseline and 3 Months
Measure: Mean (Standard Deviation); unit: Melanin Index
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Melanin Index
  Forehead | 3.8 (3.02)
  Inner Bicep | 1.4 (0.69)
  Lower Back | 0.6 (0.63)
  Inner Forearm | 1.8 (1.12)
  Outer Forearm | 4.5 (4.45)

38. Secondary Outcome: Absolute Change in Melanin Index at 6 Months Compared to Baseline
Description: as for outcome 37
Time Frame: Baseline and 6 Months
Population: Participant 005 did not have skin reflectometry measurements for any site at Month 6.
Measure: Mean (Standard Deviation); unit: Melanin Index
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Melanin Index
  Forehead | 2.2 (1.29)
  Inner Bicep | 2.7 (1.68)
  Lower Back | 3.3 (3.72)
  Inner Forearm | 2.1 (1.43)
  Outer Forearm | 4.4 (5.80)

39. Secondary Outcome: Absolute Change in Melanin Index at 9 Months Compared to Baseline
Description: as for outcome 37
Time Frame: Baseline and 9 Months
Population: Participant 002 did not have skin reflectometry measurements for any site at Month 9.
Measure: Mean (Standard Deviation); unit: Melanin Index
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Melanin Index
  Forehead | 2.4 (1.98)
  Inner Bicep | 1.9 (1.60)
  Lower Back | 3.2 (3.23)
  Inner Forearm | 2.1 (1.33)
  Outer Forearm | 2.2 (2.48)

40. Secondary Outcome: Absolute Change in Melanin Index at 12 Months Compared to Baseline
Description: as for outcome 37
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: Melanin Index
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Melanin Index
  Forehead | 3.7 (3.29)
  Inner Bicep | 2.3 (1.90)
  Lower Back | 2.0 (1.55)
  Inner Forearm | 2.2 (1.96)
  Outer Forearm | 3.4 (3.38)

41. Secondary Outcome: Percent Change in Melanin Index at 3 Months Compared to Baseline
Description: Microflash 200D is a diffuse reflectance spectrophotometer that uses a prism photodiode to provide information at 10 nm increments along the visual spectrum from 400 to 700 nm. Percent reflectance (PR) at a specific wavelength was placed into context by relating it to the reflectance of a blank at the equivalent wavelength (i.e. relating the object's reflectance to the maximum reflectance possible). Melanin (M) index was calculated as follows:
  Eqn 1= [ (PR at 650nm + PR at 660nm + 0.5*PR at 640nm + 0.5*PR at 670nm)/3 ]/100; M index = 100*log (1/Eqn 1) Higher values of M index correspond to higher melanin concentrations. Measurements were collected 5 times at each visit from each of the following sites:forehead, inner forearm, outer forearm, inner bicep and lower back. The mean of these five measurements was calculated at each visit. Percent change from baseline was calculated using these mean values.
Time Frame: Baseline and 3 Months
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Percentage change
  Forehead | 15.0 (12.90)
  Inner Bicep | 6.7 (3.50)
  Lower Back | 2.8 (3.34)
  Inner Forearm | 8.6 (5.84)
  Outer Forearm | 18.9 (19.90)

42. Secondary Outcome: Percent Change in Melanin Index at 6 Months Compared to Baseline
Description: as for outcome 41
Time Frame: Baseline and 6 Months
Population: Participant 005 did not have skin reflectometry measurements for any site at Month 6.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Percentage change
  Forehead | 8.4 (4.62)
  Inner Bicep | 12.7 (8.31)
  Lower Back | 17.0 (19.52)
  Inner Forearm | 10.2 (7.50)
  Outer Forearm | 19.2 (24.93)

43. Secondary Outcome: Percent Change in Melanin Index at 9 Months Compared to Baseline
Description: as for outcome 41
Time Frame: Baseline and 9 Months
Population: Participant 002 did not have skin reflectometry measurements for any site at Month 9.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 4
Percentage change
  Forehead | 9.2 (7.30)
  Inner Bicep | 8.9 (7.89)
  Lower Back | 15.8 (16.17)
  Inner Forearm | 9.5 (6.15)
  Outer Forearm | 8.8 (10.63)

44. Secondary Outcome: Percent Change in Melanin Index at 12 Months Compared to Baseline
Description: as for outcome 41
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Percentage change
  Forehead | 14.7 (14.11)
  Inner Bicep | 10.9 (9.43)
  Lower Back | 10.2 (7.92)
  Inner Forearm | 10.4 (10.19)
  Outer Forearm | 13.3 (13.44)

45. Secondary Outcome: Absolute Change in Electroretinogram (ERG) at Month 6 as Compared to Baseline.
Description: Amplitude for the ERG parameter, Dark Adaptation (DA) Comb B, was measured at each visit. Participants left and right eye will be analyzed.
Time Frame: Baseline and 6 months
Population: Right eyes (OD) and left eyes (OS)
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
µV
  OD: number analyzed (eyes) | 5
  OD | 38.6 (27.93)
  OS: number analyzed (eyes) | 5
  OS | 76.2 (29.06)

46. Secondary Outcome: Absolute Change in Electroretinogram (ERG) at Month 12 as Compared to Baseline.
Description: as for outcome 45
Time Frame: Baseline and 12 months
Population: Right eyes (OD) and left eyes (OS)
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Number analyzed (eyes) | 10
µV
  OD: number analyzed (eyes) | 5
  OD | 27.8 (16.66)
  OS: number analyzed (eyes) | 5
  OS | 85.8 (83.83)

47. Secondary Outcome: Qualitative Change in Hair Pigmentation at 3 Months Compared to Previous Visit.
Description: Qualitative change in hair pigmentation was measured as a binary endpoint (no change vs. increase) at Month 3 compared to previous visit.
Time Frame: Baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in hair pigmentation | 1
  Increase in hair pigmentation | 4

48. Secondary Outcome: Qualitative Change in Hair Pigmentation at 6 Months Compared to Previous Visit.
Description: Qualitative change in hair pigmentation was measured as a binary endpoint (no change vs. increase) at Month 6 compared to Month 3
Time Frame: 3 Months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in hair pigmentation | 3
  Increase in hair pigmentation | 2

49. Secondary Outcome: Qualitative Change in Hair Pigmentation at 9 Months Compared to Previous Visit.
Description: Qualitative change in hair pigmentation was measured as a binary endpoint (no change vs. increase) at Month 9 compared to Month 6
Time Frame: 6 Months and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in hair pigmentation | 4
  Increase in hair pigmentation | 1

50. Secondary Outcome: Qualitative Change in Hair Pigmentation at 12 Months Compared to Previous Visit.
Description: Qualitative change in hair pigmentation was measured as a binary endpoint (no change vs. increase) at Month 12 compared to Month 9
Time Frame: 9 Months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in hair pigmentation | 5
  Increase in hair pigmentation | 0

51. Secondary Outcome: Qualitative Change in Skin Pigmentation at 3 Months Compared to Previous Visit.
Description: Qualitative change in skin pigmentation was measured as a binary endpoint (no change vs. increase) at Month 3 compared to previous visit.
Time Frame: Baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in skin pigmentation | 4
  Increase in skin pigmentation | 1

52. Secondary Outcome: Qualitative Change in Skin Pigmentation at 6 Months Compared to Previous Visit.
Description: Qualitative change in skin pigmentation was measured as a binary endpoint (no change vs. increase) at Month 6 compared to Month 3
Time Frame: 3 Months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in skin pigmentation | 5
  Increase in skin pigmentation | 0

53. Secondary Outcome: Qualitative Change in Skin Pigmentation at 9 Months Compared to Previous Visit.
Description: Qualitative change in skin pigmentation was measured as a binary endpoint (no change vs. increase) at Month 9 compared to Month 6
Time Frame: 6 Months and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in skin pigmentation | 5
  Increase in skin pigmentation | 0

54. Secondary Outcome: Qualitative Change in Skin Pigmentation at 12 Months Compared to Previous Visit.
Description: Qualitative change in skin pigmentation was measured as a binary endpoint (no change vs. increase) at Month 12 compared to Month 9
Time Frame: 9 Months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in skin pigmentation | 5
  Increase in skin pigmentation | 0

55. Secondary Outcome: Qualitative Change in Fundus Pigmentation at 3 Months Compared to Previous Visit.
Description: Qualitative change in fundus pigmentation was measured as a binary endpoint (no change vs. increase) at Month 3 compared to previous visit.
Time Frame: Baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in fundus pigmentation | 5
  Increase in fundus pigmentation | 0

56. Secondary Outcome: Qualitative Change in Fundus Pigmentation at 6 Months Compared to Previous Visit.
Description: Qualitative change in fundus pigmentation was measured as a binary endpoint (no change vs. increase) at Month 6 compared to Month 3
Time Frame: 3 Months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in fundus pigmentation | 5
  Increase in fundus pigmentation | 0

57. Secondary Outcome: Qualitative Change in Fundus Pigmentation at 9 Months Compared to Previous Visit.
Description: Qualitative change in fundus pigmentation was measured as a binary endpoint (no change vs. increase) at Month 9 compared to Month 6
Time Frame: 6 Months and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in fundus pigmentation | 5
  Increase in fundus pigmentation | 0

58. Secondary Outcome: Qualitative Change in Fundus Pigmentation at 12 Months Compared to Previous Visit.
Description: Qualitative change in fundus pigmentation was measured as a binary endpoint (no change vs. increase) at Month 12 compared to Month 9
Time Frame: 9 Months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
Participants
  No change in fundus pigmentation | 5
  Increase in fundus pigmentation | 0

59. Secondary Outcome: Absolute Change in Hair Melanin at 12 Months Compared to Baseline
Description: Hair melanin was assessed using pyrrole-2,3,5-tricarboxylic acid (PTCA), a marker of eumelanin and 4-amino-3-hydroxyphenylalanine (4-AHP), a marker of pheomelanin.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
ng/mg
  PTCA | 8.38 (5.11)
  4-AHP | 5.92 (11.68)

60. Secondary Outcome: Percent Change in Hair Melanin at 12 Months Compared to Baseline
Description: as for outcome 59
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
percentage change
  PTCA | 50.30 (45.92)
  4-AHP | 27.23 (23.22)

61. Other Pre Specified Outcome: Number of Ocular Adverse Events
Time Frame: Study duration, up to 18 months
Measure: Number; unit: ocular adverse events
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
ocular adverse events | 0

62. Other Pre Specified Outcome: Number of Non-ocular Adverse Events
Time Frame: Study duration, up to 18 months
Measure: Number; unit: non-ocular adverse events
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
non-ocular adverse events | 10

63. Other Pre Specified Outcome: Severity of Adverse Events
Time Frame: Study duration, up to 18 months
Measure: Number; unit: adverse events
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
adverse events
  Mild | 9
  Moderate | 1

64. Other Pre Specified Outcome: Number of Adverse Events Related to Investigational Product (IP)
Time Frame: Study duration, up to 18 months
Measure: Number; unit: adverse events related to IP
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
adverse events related to IP | 0

65. Other Pre Specified Outcome: Number of Participants Withdrawn From Investigational Product (IP) Due to Safety and Abnormal Laboratory Results
Time Frame: Study duration, up to 18 months
Measure: Number; unit: participant withdrawals
Arm/Group | Nitisinone
Number analyzed (Participants) | 5
participant withdrawals | 0

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: Adverse events were collected on and after the baseline visit, and when investigational product (IP) began.
Arm/Group | Nitisinone
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitisinone (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemangioma (Vascular disorders) | 1 (1)
Neurological examination abnormal (Investigations) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes